CLINICAL TRIAL: NCT00004077
Title: A Study of Paclitaxel, Cisplatin and Ifosfamide as Induction Therapy in the Treatment of Patients Relapsing After BEP Chemotherapy for Metastatic Germ Cell Tumors
Brief Title: Paclitaxel, Ifosfamide, and Cisplatin in Treating Patients With Metastatic Testicular Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067286; MRC-TIP; EU-99012
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-01

CONDITIONS: Testicular Germ Cell Tumor
Keywords: stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and yolk sac tumor; testicular yolk sac tumor and teratoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Carcinoma, Embryonal | interventions — Cisplatin; Ifosfamide; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel, ifosfamide, and cisplatin in treating patients who have metastatic testicular cancer that has recurred following treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of combining paclitaxel, ifosfamide, and cisplatin induction in patients with metastatic nonseminomatous germ cell tumor of the testis in first relapse following first line treatment with bleomycin, etoposide, and cisplatin.
* Determine the response rates to this regimen in these patients

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours and ifosfamide IV and cisplatin IV daily for 5 days. Patients with stable or responding disease repeat treatment every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A minimum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Metastatic nonseminomatous germ cell tumor of the testis

  * In first relapse following first line treatment with bleomycin, etoposide, and cisplatin
  * Biopsy proven germ cell tumor OR
  * Rising tumor markers (alpha fetoprotein and/or human chorionic gonadotropin)
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 16 to 64

Performance status:

* 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Glomerular filtration rate greater than 50 mL/min

Other:

* No other prior malignancy except curatively treated nonmelanomatous skin cancer or superficial bladder cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior experimental drugs

Ages: 16 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 1996-05; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm D. Mason, MD, Study Chair — Velindre NHS Trust
Locations (1):
- Velindre Hospital, Cardiff, Wales, United Kingdom

REFERENCES:
- [Result] Mead GM, Cullen MH, Huddart R, Harper P, Rustin GJ, Cook PA, Stenning SP, Mason M; MRC Testicular Tumour Working Party. A phase II trial of TIP (paclitaxel, ifosfamide and cisplatin) given as second-line (post-BEP) salvage chemotherapy for patients with metastatic germ cell cancer: a medical research council trial. Br J Cancer. 2005 Jul 25;93(2):178-84. doi: 10.1038/sj.bjc.6602682. PMID 15999102